CLINICAL TRIAL: NCT02894983
Title: Comparison of Volar-flexion, Ulnar-deviation and Functional Position Cast Immobilization in the Non-operative Treatment of Distal Radius Fracture in Elderly Patients: a Pragmatic Randomized Controlled Trial
Brief Title: Conservative Treatment of Distal Radius Fracture in Elderly in Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Central Finland Hospital District (Other); Satakunta Central Hospital (Other)
Responsible Party: Principal Investigator, Teemu Hevonkorpi, MBBS, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R16035
Record Dates: First submitted 2016-08-22; First posted 2016-09-09 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Colles' Fracture; Distal Radius Fracture
Keywords: wrist fracture; colles fracture; non-operative; rehabilitation
MeSH Terms: conditions — Colles' Fracture; Wrist Fractures | interventions — Conservative Treatment

ARMS (2):
- Arm 1 (Other): Conservative treatment chosen by physician on-call for dorsally displaced radius fracture.
  Interventions: Other: Flexion-ulnar cast
- Arm 2 (Other): Conservative treatment chosen by physician on-call for dorsally displaced radius fracture.
  Interventions: Other: Functional cast

INTERVENTIONS:
Other: Flexion-ulnar cast — The group will be treated with closed reduction and flexion-ulnar deviation position cast. This will take place under local anaesthesia by means of local infiltration commonly used in Finland. There is no preferable method for performing the reduction. Additional radiographs will be taken to verify the success of the reduction one week after the reduction and after two and five weeks of casting if treating health care professional it requires. The cast will be disposed after 5 weeks.
  Other Names: Conservative treatment
  Arms: Arm 1
Other: Functional cast — The group will be treated with closed reduction and functional position cast. This will take place under local anaesthesia by means of local infiltration commonly used in Finland. There is no preferable method for performing the reduction. Additional radiographs will be taken to verify the success of the reduction one week after the reduction and after two and five weeks of casting if treating health care professional it requires. The cast will be disposed after 5 weeks.
  Other Names: Conservative treatment
  Arms: Arm 2

SUMMARY:
There is no consensus about the best conservative treatment for patients with dorsally displaced distal radius fractures. The previous studies that have examined the most valid method for cast immobilization have lacked uniform and patient-rated outcome measures, proper randomization and sufficient study population. The aim of this study is to compare functional position cast to flexion-ulnar -deviation with dorsally displaced distal radius fractures in patients aged 65 years or older. The conservative treatment is performed in clinical practice by various health care professionals with different techniques of reduction which are not limited to any specific technique in this pragmatic, randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Low energy intra- or extra-articular dorsal primarily stable, reducible DRF within 3 cm of the radiocarpal joint diagnosed with lateral and posterior-anterior radiographs in ER
* Physician on-call (general practitioner, acute physician, orthopedic resident, orthopedic consult) thinks patient could be appropriate for non-operative treatment

Exclusion Criteria:

* Operative treatment
* Refuse to participate the study
* Open fracture more than Gustilo 1 gradus
* Age under 65 years
* Chauffeure's or Barton´s fracture
* Smith´s fracture (volar angulation of the fracture)
* Does not understand written and spoken guidance in local languages
* Pathological fracture or previous fracture in the same wrist, forearm or elbow

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 114 (Actual)
Dates: Start 2016-06; Primary Completion 2018-04 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Patient Rated Wrist Evaluation (PRWE) measure is the primary outcome measure of wrist pain and disability in the study | 2 years
  The PRWE comprises 15 questions to measure wrist pain and disability in daily activities. In PRWE patients rate wrist pain and disability from 0 to 10 and it consists three subscales: Pain, Function and Cosmetics.

SECONDARY OUTCOMES:
Disability of the wrist measured with the Disability of the Arm, Shoulder and Hand (QuickDASH) questionnaire. | 2 years
  The QuickDASH is self-reported questionnaire and shortened version of DASH outcome measure to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb in 11 dimensions in 1-5 scale.
Quality of life measured with the 15-D. | 2 years
  The 15D is a validated, generic, self-administered instrument for assessing the health related quality of life among adults. It combines the advantages of a preference-based and single index measure on a 0-1 scale.
Pain measured in Visual Analogue Scale (VAS). | Baseline, 3 months, 1 year, 2 years
  The VAS is derived by health care professional question of pain in scale 0 to 10 in which 0 implies no pain and 10 the worst possible pain.
Range of motion (ROM) is measured with a goniometer | 3 months
  The ROM of the wrist is measured on both hands with a handheld goniometer in degrees.
Grip strength is measured with a dynamometer | 3 months
  Grip strength is measured with a dynamometer in kg as the mean of three measurements. It will be numbered in percentage of the uninjured side.
The pain catastrophizing scale (PCS) is measured with a self-administered questionnaire. | 2 years
  The PCS is designed to measure person's willingness to catastrophize the pain while they are experiencing it. In the questionnaire patients answer questions about how they feel and think when they are in pain and it can be taken while they are not experiencing pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ville Mattila, MD, Professor, Study Director — Tampere Univeristy Hospital; Antti Launonen, MD, PhD, Principal Investigator — Tampere University Hospital; Teemu Hevonkorpi, MBBS, Study Chair — Tampere University Hospital; Lauri Raittio, MBBS, Study Chair — Tampere University Hospital; Toni Luokkala, MD, Study Chair — Central Finland Central Hospital; Aleksi Reito, MD, PhD, Study Chair — Central Finland Central Hospital; Juha Kukkonen, MD, PhD, Study Chair — Satakunta Central Hospital; Minna Laitinen, Adjacent prof, Study Chair — Tampere University Hospital
Locations (3):
- Finland (3):
  - Central Finland Central Hospital, Jyväskylä
  - Satakunta Central Hospital, Pori
  - Tampere Univeristy Hospital, Tampere

REFERENCES:
- [Derived] Ax M, Reito A, Hevonkorpi TP, Palola V, Kukkonen J, Luokkala T, Laitinen MK, Launonen AP, Mattila VM. A comparison of the functional results and costs of functional cast and volar-flexion ulnar deviation cast at 2-year follow-up in 105 patients aged 65 and older with dorsally displaced distal radius fracture: A randomized controlled trial. PLoS One. 2023 Apr 6;18(4):e0283946. doi: 10.1371/journal.pone.0283946. eCollection 2023. PMID 37023069
- [Derived] Raittio L, Launonen AP, Hevonkorpi T, Luokkala T, Kukkonen J, Reito A, Laitinen MK, Mattila VM. Two casting methods compared in patients with Colles' fracture: A pragmatic, randomized controlled trial. PLoS One. 2020 May 29;15(5):e0232153. doi: 10.1371/journal.pone.0232153. eCollection 2020. PMID 32469881
- [Derived] Raittio L, Launonen A, Hevonkorpi T, Luokkala T, Kukkonen J, Reito A, Sumrein B, Laitinen M, Mattila VM. Comparison of volar-flexion, ulnar-deviation and functional position cast immobilization in the non-operative treatment of distal radius fracture in elderly patients: a pragmatic randomized controlled trial study protocol. BMC Musculoskelet Disord. 2017 Sep 18;18(1):401. doi: 10.1186/s12891-017-1759-y. PMID 28923035